CLINICAL TRIAL: NCT01478061
Title: Multi-center Assessment of Grafts in Coronaries: Long-term Evaluation of the C-Port Device
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardica, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2007-01
Record Dates: First submitted 2011-10-19; First posted 2011-11-23 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases | interventions — Anastomosis, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anastomoses in blood vessels and grafts (Active Comparator)
  Interventions: Device: Anastomosis (C-Port® )

INTERVENTIONS:
Device: Anastomosis (C-Port® ) — creation of anastomoses in blood vessels and grafts, including use in coronary artery bypass grafting procedures
  Other Names: C-Port® Distal Anastomosis System; C-Port® xA™ Distal Anastomosis System; C-Port® FlexA™ Distal Anastomosis System; C-Port® XCHANGE™ Distal Anastomosis System

SUMMARY:
The Study plan is a post-market prospective, multi-center, open-label registry. The vein graft failure rates for the currently commercialized C-Port devices will be compared to an a priori rate taken from the peer-reviewed literature.

DETAILED DESCRIPTION:
To satisfy the requirements set forth in post-market surveillance orders issued by the US FDA to Cardica, Inc., the following outcomes will be evaluated:

1. Acute, midterm, and one-year graft failure rates for coronary revascularization using the C-Port® xA™ Distal Anastomosis System, C-Port® FlexA™ Distal Anastomosis System, and C-Port® XCHANGE™ Distal Anastomosis System when in general use in the United States compared to hand-sewn anastomoses.
2. Technical failure rates when attempting to complete an anastomosis using the C-Port xA, FlexA, and XCHANGE Distal Anastomosis Systems.
3. The technical success rate of hand-sewn anastomoses following technical failures of the C-Port devices and the hand-sewn graft patency rates and clinical sequelae at one year.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent.
* Willing and able to have follow-up visits and examinations.
* Less than 80 years old.
* Have an ejection fraction of >30 %.
* Have a life expectancy of >1 year.

Pre-Operative Exclusion Criteria:

* Currently participating in other clinical trials that would conflict with this protocol.
* Unable to meet study requirements.
* Currently pregnant.
* Require preoperative use of an intraaortic balloon pump.
* Have a history of a bleeding disorder or history of a thromboembolic disease requiring anticoagulation therapy.
* Have congestive heart failure or been classified as NYHA Class IV.
* Have an aspirin allergy or other contraindications to aspirin use.
* Previous coronary artery bypass surgery.
* Vasculitis or other nonatherosclerotic cause for coronary artery disease.

Intra-Operative Exclusion Criteria:

* At least one target vessel site where the C-Port anastomosis will be placed that is free from severe calcification or severe atheromas
* Target vessel wall properties where the C-Port anastomosis will be placed are suitable for hand-sewn anastomosis
* Target vessel diameter is ≥ 1.3 mm
* Target vessel has a single wall thickness ≤ 0.75mm
* Hemodynamically stable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Graft patency rates for coronary revascularization when in general use in the United States compared to hand-sewn anastomoses. | 12 months
  a. Acute, midterm, and one-year graft patency rates for coronary revascularization when in general use in the United States compared to hand-sewn anastomoses.

SECONDARY OUTCOMES:
Technical Failure Rates | Day 1
  Technical failure rates when completing an anastomosis using the C-Port products.
Technical success rate of hand-sewn | Day 1 and 12 months
  The technical success rate of hand-sewn anastomoses following technical failures of the C-Port products and the hand-sewn graft patency rates and clinical sequelae at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Husam Balkhy, MD, Principal Investigator — Wisconsin Heart Hospital
Locations (7):
- United States (7):
  - University of Arkansas, Little Rock, Arkansas
  - Genesis Medical Center, Davenport, Iowa
  - Lenox Hill Hospital, New York, New York
  - Akron General Medical Center, Akron, Ohio
  - Cardiopulmonary Research Science & Technology Institute, Dallas, Texas
  - Methodist Hospital - Houston, Houston, Texas
  - Wisconsin Heart, Wauwatosa, Wisconsin